CLINICAL TRIAL: NCT02819882
Title: A Prospective Registry Study in Patients With Unresectable Locally Advanced or Metastatic Breast Cancer (MBC)
Acronym: REGISTEM
Status: Recruiting | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Hoffmann-La Roche (Industry); Novartis (Industry); AstraZeneca (Industry); Pfizer (Industry); Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: GEICAM 2014-03
Record Dates: First submitted 2016-06-20; First posted 2016-06-30 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasms
Keywords: Unresectable; locally; advanced; metastatic disease
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood samples Primary and metastatic lesion tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Luminal A-like subtype: Patients that express Estrogen receptor (ER), express Progesterone Receptor (PgR)+ (≥ 20%), don't express HER2 and have Ki-67 'low' (< 14%).
  Interventions: Other: No intervention
- Luminal B-like (HER2 negative) subtype:: Patients that express ER and are either PgR- or low (< 20%) and/or Ki67 'high' (≥ 14%).
  Interventions: Other: No intervention
- Luminal B-like (HER2 positive) subtype:: Patients that express ER and HER2 irrespective of PgR or Ki67 status.
  Interventions: Other: No intervention
- HER2-enriched subtype: Patients that express HER2 and don't express ER or PgR.
  Interventions: Other: No intervention
- Triple Negative (TN) subtype: Patients who are negative for the expression of ER, PgR and HER2.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This study is a prospective, multicenter non-interventional cohort study designed to develop a registry in unresectable locally advanced or metastatic disease.

DETAILED DESCRIPTION:
The target population for inclusion in this study is breast cancer patients recently diagnosed (from January 2016) with unresectable locally advanced or metastatic disease (either after a recurrence or as first diagnosis). No treatment regimen will be protocol specified. This is an observational study in which clinical decisions concerning the optimum management strategy for a particular patient are taken independently of and/or prior to, any decision by the physician to invite a patient to participate in the study. The treating physician will make all treatment decisions according to his/her regular clinical practice independent of this study. Patients enrolled on the study are free to withdraw their informed consent for the use and disclosure of health information at any time and when asked, patients are not obliged to provide a reason. Patients may request discontinuation from the study at any time.

The date and the reason for withdrawal or discontinuation from the study must be recorded in the electronic case report form (eCRF). An attempt will be made to determine the date of discontinuation and final status (i. e. withdrawal of consent, loss to follow-up, death) of any patient who discontinues from the study. However, the treating clinician is encouraged to follow the patient as long as possible, until patient death or through study end. The Sponsor has the right to terminate the study at any time. The Sponsor will notify the investigator if the study is placed on hold or if the Sponsor decides to discontinue the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (males or females) diagnosed with unresectable locally advanced or MBC (either after a recurrence or as first diagnosis) from January 2016 onwards.
2. Patients who died are allowed to be included on the study.
3. Able and willing to provide written informed consent if they are alive.
4. Age ≥ 18 years.
5. Availability to medical records access and all data related to the disease management.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for inclusion in this study is breast cancer patients recently diagnosed (from January 2016) with unresectable locally advanced or metastatic disease (either after a recurrence or as first diagnosis).
Sampling Method: Non-Probability Sample
Enrollment: 1867 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with the different breast cancer subtypes and real distribution of them. | 8 years
  Number of patients with the different breast cancer subtypes (Luminal A-like, Luminal B-like [HER2 negative], Luminal B-like [HER2 positive], HER2-enriched and Triple Negative) of the unresectable locally advanced or metastatic disease

SECONDARY OUTCOMES:
Patient and tumor characteristics and frequency of breast cancer with heredofamiliar risk. | 8 years
  It will be performed a table with patient and tumor characteristics including only those patients with heredofamiliar risk.
Differences in the development disease in the group of male vs female patients. | 8 years
  It will be performed an analysis separately for each subtype and by male and female and it will analyse if there are any significative difference between them.
Influence of timing of primary tumor surgery in patients with metastatic disease as first diagnosis | 8 years
  Influence of timing of primary tumor surgery in patients with metastatic disease as first diagnosis
Number of participants with specific biomarkers on tumor and blood samples. | 8 years
  to improve the understanding of metastatic breast cancer by performing analysis on tumor and blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Study Director, Study Director — Hospital de Donostia, San Sebastián, Spain; Study Director, Study Director — Hospital Universitario Gregorio Marañón, Madrid, Spain; Study Director, Study Director — Instituto Valenciano de Oncología (IVO), Valencia, Spain; Study Director, Study Director — Complejo Hospital Universitario A Coruña (CHUAC), Galicia, Spain; Study Director, Study Director — Hospital Universitario Fundación Jimenez Díaz, Madrid, Spain
Locations (40):
- Spain (40):
  - Hospital General de Elche, Elche, Alicante
  - Althaia-Xarxa Assistencial de Manresa, Manresa, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Hospital Universitario Donostia, San Sebastián, Donostia
  - Hospital Dr. Negrín, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Infanta Sofía, San Sebastián de los Reyes, Madrid
  - Hospital Son Llatzer, Palma de Mallorca, Mallorca
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital Universitario de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital San Juan de Alicante, Alicante
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - ICO L´Hospitalet, Barcelona
  - Hospital Universitario Germans Trias i Pujol, Barcelona
  - Hospital Moisés Broggi_institut Catalá D´Oncologia, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital de León, León
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario de Málaga, Málaga
  - Hospital Clínico Universitario Virgen de la Arrixaca, Murcia
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - IVO-Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hosital General de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org